CLINICAL TRIAL: NCT06808191
Title: Effect of Magnetic Current on Chronic Ulcer Healing of Diabetic Foot
Brief Title: Effect of Magnetic Current on Ulcer Healing
Acronym: ulcer healing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mahmoud Awad Ramadan Elkholy, lecturer of physical therapy for integumentary system disorders, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/03032024/Kamel
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: ulcer diabetic magnetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: diabetic patients (n=40) affected with diabetic foot ulcer(s) will be recruited in the study and will be randomly allocated into two equal groups (20 patients in each group):
  1. Group A: Pulsed electromagnetic field (PEMF) group.
  2. Group B: Control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): Pulsed electromagnetic therapy will be delivered at the frequency of 12Hz, with magnetic flux density of 12G. Each treatment session will last for 1 hour, which will be repeated for 14 sessions within 3weeks. 20 patients will remain in the study until the wound heals or 14 sessions will be completed, whichever came first
  Interventions: Device: pulsed electromagnetic currant machine
- Group B (Placebo Comparator): 20 patients will receive intervention by using the same PEMF unit, but the output will be shut off.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: pulsed electromagnetic currant machine — Pulsed electromagnetic therapy will be delivered at the frequency of 12Hz, with magnetic flux density of 12G. Each treatment session will last for 1 hour, which will be repeated for 14 sessions within 4weeks.
  Arms: group A
Other: Placebo — control group will receive intervention by using the same PEMF unit, but the output will be shut off.
  Arms: Group B

SUMMARY:
This study aims to evaluate the effectiveness of magnetic current in the management of DFUs as an alternative therapy on promoting the healing of chronic diabetic foot ulcers as compared with a control group.Twenty diabetic patients (n=40) affected with diabetic foot ulcer(s) will be recruited in the study and will be randomly allocated into two equal groups (20 patients in each group):

1- Group A: Pulsed electromagnetic field (PEMF) group. 2- Group B: Control group. Assessments of the healing of ulcers will be performed at the baseline, post-treatment evaluation (ie, after 14 treatment sessions), and 1-month follow-up.

:

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of magnetic current in the management of DFUs as an alternative therapy on promoting the healing of chronic diabetic foot ulcers as compared with a control group.Twenty diabetic patients (n=40) affected with diabetic foot ulcer(s) will be recruited in the study and will be randomly allocated into two equal groups (20 patients in each group):

1. Group A: Pulsed electromagnetic field (PEMF) group.
2. Group B: Control group. Assessments of the healing of ulcers will be performed at the baseline, post-treatment evaluation (ie, after 14 treatment sessions), and 1-month follow-up.

Outcome measures will include:

1. Wound closure.
2. Wound depth.
3. Microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* 1. The ankle brachial index should fall between 0.9 and 1.2 to reassure that arterial insufficiency was not causing or contributing to the nonhealing wound.

  2. Patients diagnosed with diabetes with unsatisfactory healing of ulcer(s) in the preceding 4 weeks.

  3. Wagner grade 1 or 2 ulcers on the foot without exposure of bone, muscle, ligaments, or tendons.

Exclusion Criteria:

- 1- Ulcers secondary to non-diabetic etiology. 2- Poorly controlled diabetes. 3- Pregnancy. 4- Patients wearing a pacemaker or with malignancy or history of radiotherapy. 5- Patients who were taking medications that might affect their circulation or sensation and motor functioning and patients with any history of alcoholism were also excluded.

6- Patients who had clinical signs of infection or were taking antibiotics at the time of enrollment.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
ulcer size | 4 weeks
  smart phone applications used to calculate wound size
Doppler ultrasonography | 4 weeks
  used to calculate wound depth and microcirculation angiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: heba mohamed ali, Professor of Physical therapy, Study Chair — beni suif university; mahmoud awd elkholy, lecturer of physical therapy, Study Director — beni suif university; asmaa ramadan kamel, physiotherapist, Principal Investigator — beni suif university
Locations (1):
- Beni-Suif University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i dont know

REFERENCES:
- [Background] Kwan RL, Cheing GL, Vong SK, Lo SK. Electrophysical therapy for managing diabetic foot ulcers: a systematic review. Int Wound J. 2013 Apr;10(2):121-31. doi: 10.1111/j.1742-481X.2012.01085.x. Epub 2012 Sep 7. PMID 22958779